CLINICAL TRIAL: NCT01759992
Title: Determination of the Effects and Costs of Respiratory Muscle Training in Institutionalized Elderly People With Functional Impairment: A Randomized Controlled Trial
Brief Title: Effects and Costs of Respiratory Muscle Training in Institutionalized Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Maria dels Angels Cebria i Iranzo, PT, PhD, Assistant Professor, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UV-INV-PRECOMP12-80293; H1335803152705 (Other: University of Valencia Research Ethics Committee)
Record Dates: First submitted 2012-12-31; First posted 2013-01-03 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Muscle Weakness; Syndrome; Institutionalization; Respiratory Morbidity; Cardiovascular Morbidity
Keywords: Frail elderly; Muscle weakness; Institutionalization; Respiratory muscle training
MeSH Terms: conditions — Muscle Weakness; Syndrome | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Usual care
- Treatment group (Experimental): Participants will breathe against a load ≥ 50% of their baseline MIP, after which loads will increase according to the participant's tolerance across the remaining training period, using a Borg scale rating of 4 to 6 on perceived exertion as an indicator of adequate training intensity.
  Interventions: Device: Threshold® Inspiratory Muscle Trainer (treatment).

INTERVENTIONS:
Device: Threshold® Inspiratory Muscle Trainer (treatment). — Interval-based program consisting of seven cycles of 2-minutes work and 1-minute rest. The sessions will take place 3 times per week over a eight-week period for a total of 24 sessions. All participants were familiarized with the breathing exercises over a two-week familiarization period at the beginning of the protocol. The load will be adjusted at ≥ 50% of baseline MIP.
  Other Names: Respironics® Health Scan Inc. Cedar Grove, NJ, USA
  Arms: Treatment group

SUMMARY:
The global loss of muscle mass and strength associated with aging is a cause of functional impairment and disability, particularly in the older elderly (>80 years). Respiratory function can be severely compromised if there is a decrease of respiratory (RM) strength complicated by the presence of comorbidities and physical immobility. In this context, the need for supportive services involves the need for long-term care and consequently the institutionalization.

Previous studies have shown that the increase of RM strength has positive healthy effects, such as the increase in functional capacity, the decrease in RM fatigue, the decrease of dyspnoea and the improvement of quality of life, both in healthy people and patients. Therefore, specific RM training may be regarded as a beneficial alternative to improve RM function, and thus prevent physical and clinical deterioration in this frail population.

Study hypothesis: The inspiratory muscle training (IMT) would improve respiratory muscle strength and endurance, exercise capacity and quality of life in an elderly population, who are unable to engage in general exercise conditioning.

ELIGIBILITY:
Inclusion Criteria:

* People aged > 65 years
* Barthel Index < 75 score
* Mini-mental state examination ≥ 20 score
* Inspiratory muscle weakness (MIP ≤ 30% predicted value)

Exclusion Criteria:

* Ability to independently walk more than 14 m
* Significant chronic cardiorespiratory diagnoses
* Acute cardiorespiratory episode during the 2 previous months
* Neurological, muscular, or neuromuscular problems interfering with the capacity to engage in the tests and training protocol
* Active smokers or former smokers (< 5 years)
* A terminal disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximum Inspiratory Pressure (MIP) | The groups were assessed at baseline (time zero) and at the end of the training protocol (week 9).
  MIP is probably the most frequently reported noninvasive estimates of inspiratory muscle strength. Ever since Black and Hyatt (1969) reported this technique it has been widely used in patients, healthy control subjects across all ages, and athletes. Pressure is recorded at the mouth during a quasi-static short (few seconds) maximal inspiration. The manoeuvre is generally performed at Residual Volume (RV). Reference: Am J Respir Crit Care Med. 2002;166:531-535.
Maximum Expiratory Pressure (MEP) | The groups were assessed at baseline (time zero) and at the end of the training protocol (week 9).
  MEP is probably the most frequently reported noninvasive estimates of expiratory muscle strength. Ever since Black and Hyatt (1969) reported this technique it has been widely used in patients, healthy control subjects across all ages, and athletes. Pressure is recorded at the mouth during a quasi-static short (few seconds) maximal expiration. The manoeuvre is generally performed at Total Lung Capacity (TLC). Reference: Am J Respir Crit Care Med. 2002;166:531-535.

SECONDARY OUTCOMES:
Maximal Voluntary Ventilation (MVV) | The groups were assessed at baseline (time zero) and at the end of the training protocol (week 9).
  This ventilatory test is a non-invasive technique and is a measure of both inspiratory and expiratory muscle endurance. The MVV is the largest volume that can be breathed in and out of the lungs during a 12 -15 second interval with maximal voluntary effort. Reference: Am J Respir Crit Care Med. 2002;166:562-564.
Time performed to walk 10 m distance (10mWT). | The groups were assessed at baseline (time zero) and at the end of the training protocol (week 9).
  The 10-Meter Walk Test (10mWT) is a measure of gait speed. The walking course consist of 14 m in a hallway: a 2 m warm-up, 10 m use for the speed measurement, and 2 m for slowing down to stop. Participants can use the assistive device (eg, cane, walker) or orthotic device (eg, ankle-foot orthosis) that they use "most often" (if any) at each time point. Reference: Tilson JK, Sullivan KJ, Cen SY, et al. Meaningful gait speed improvement during the first 60 days poststroke: minimal clinically important difference. Phys Ther. 2010;90(2):196-208.
Maximal heart rate achieved at the end of the incremental arm ergometry test. | The groups were assessed at baseline (time zero) and at the end of the training protocol (week 9).
  The incremental arm ergometry test begins with a 3 minutes warm-up (50-70 rpm) and continues with an incremental power of 10 W each 2 minutes. The test concludes when the heart rate achieves 80% of maximum theoretical heart rate (220-age) and/or inability to maintain 50 rpm. Reference: Franklin BA. Exercise testing, training, and arm ergometry. Sports Med. 1985;2(2):100-19

OTHER OUTCOMES:
Health-related quality-of-life (CRQ). | The groups were assessed at baseline (time zero) and at the end of the training protocol (week 9).
  Chronic Respiratory Questionnaire (CRQ) is an designed instrument to evaluate the impact of interventions, including respiratory rehabilitation. The CRQ includes 20 items divided into four domains: dyspnoea (five items); fatigue (four items); emotional function (seven items); and mastery, a domain which explores how patients cope with their chronic illness (four items). Reference: Güell R, Casan P, Sangenís M, et al. Quality of life in patients with chronic respiratory disease: the Spanish version of the Chronic Respiratory Questionnaire (CRQ). Eur Respir J. 1998; 11(1):55-60.

CONTACTS AND LOCATIONS:
Overall Officials: M. Àngels Cebrià i Iranzo, PT, PhD, Principal Investigator — University of Valencia; M. Ángeles Tortosa Chuliá, PhD, Study Chair — University of Valencia; Celedonia Igual Camacho, PT, PhD, Study Chair — University of Valencia; Laura López Bueno, PT, PhD, Study Chair — University of Valencia
Locations (1):
- Grupo Gero Residencias "La Saleta", Valencia, Valencia, Spain

REFERENCES:
- [Background] Geddes EL, O'Brien K, Reid WD, Brooks D, Crowe J. Inspiratory muscle training in adults with chronic obstructive pulmonary disease: an update of a systematic review. Respir Med. 2008 Dec;102(12):1715-29. doi: 10.1016/j.rmed.2008.07.005. Epub 2008 Aug 15. PMID 18708282
- [Background] Gorzoni ML, Pires SL. [Long-term care elderly residents in general hospitals]. Rev Saude Publica. 2006 Dec;40(6):1124-30. doi: 10.1590/s0034-89102006000700024. Portuguese. PMID 17173173
- [Background] Gosselink R, De Vos J, van den Heuvel SP, Segers J, Decramer M, Kwakkel G. Impact of inspiratory muscle training in patients with COPD: what is the evidence? Eur Respir J. 2011 Feb;37(2):416-25. doi: 10.1183/09031936.00031810. PMID 21282809
- [Background] Rydwik E, Frandin K, Akner G. Physical training in institutionalized elderly people with multiple diagnoses--a controlled pilot study. Arch Gerontol Geriatr. 2005 Jan-Feb;40(1):29-44. doi: 10.1016/j.archger.2004.05.009. PMID 15531021
- [Background] Simoes RP, Castello V, Auad MA, Dionisio J, Mazzonetto M. Prevalence of reduced respiratory muscle strength in institutionalized elderly people. Sao Paulo Med J. 2009 May;127(2):78-83. doi: 10.1590/s1516-31802009000200005. PMID 19597682
- [Background] Watsford M, Murphy A. The effects of respiratory-muscle training on exercise in older women. J Aging Phys Act. 2008 Jul;16(3):245-60. doi: 10.1123/japa.16.3.245. PMID 18660549